CLINICAL TRIAL: NCT03252834
Title: To Study the Individual Variants of Chemotherapy-induced Abnormal Thermal Sensation in Cancer Patients
Brief Title: Genetic Variants and Chemotherapy-induced Abnormal Thermal Sensation
Status: Terminated | Type: Observational
Why Stopped: Poor enrollment
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Meng-Ru Shen, Associate Dean for Research, National Cheng-Kung University Hospital
Other Study IDs: B-ER-106-120
Record Dates: First submitted 2017-08-15; First posted 2017-08-17 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Chemotherapy-induced Abnormal Thermal Sensation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with endometrial or ovarian cancer
  Interventions: Diagnostic Test: Genetic variants of TRPV1, TRPM2, TRPA1 and ORAI
- Patients with colorectal cancer
  Interventions: Diagnostic Test: Genetic variants of TRPV1, TRPM2, TRPA1 and ORAI

INTERVENTIONS:
Diagnostic Test: Genetic variants of TRPV1, TRPM2, TRPA1 and ORAI — Genetic variants of TRPV1, TRPM2, TRPA1 and ORAI1 will be analyzed. Quantitative Sensory Test, QST, will be used to determined if there is abnormal thermal sensation.

SUMMARY:
This is a prospective, single arm, single center study evaluating the use of a 4-gene panel to predict the occurrence of chemotherapy-induced abnormal thermal threshold in endometrial and ovarian cancer patients receiving post-operative chemotherapy with Carboplatin/Paclitaxel, and stage III colorectal cancer patients receiving adjuvant chemotherapy with mFOLFOX6. A total of 100 patients will be enrolled during 2017 July~ 2019 June. Blood sample will be collected before chemotherapy to analyze the genetic variants of TRPV1, TRPM2, TRPA1 and ORAI1. All patients will receive neurologic examination (Quantitative Sensory Test, QST) and complete the questionnaires for quality of life (EQ5D & CIPN20). The primary endpoint of this study is to test if the genetic variant of TRPV1, TRPM2, TRPA1, and ORAI1 is a predictive biomarker for the chemotherapy-induced abnormal thermal sensation in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years old
* Pathological stage I~IV for ovarian cancer, stage II~IV for endometrial cancer, or stage III for colorectal cancer.
* Scheduled to receive adjuvant Paclitaxel/Carboplatin for ovarian or endometrial cancer, or mFOLFOX6 for colorectal cancer.
* Patient willing to provide blood sample for research purposes.
* Ability of the patient to provide informed consent.

Exclusion Criteria:

* Prior treatment with neurotoxic chemotherapy, such as oxaliplatin, cisplatin, carboplatin, taxanes or vinca alkaloids.
* Receiving chemotherapy within 6 months.
* A family history of a genetic or familial neuropathy
* Poor compliance

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Colorectal, endometrial, or ovarian cancer patients who are scheduled to receive post-operative adjuvant chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
The change of thermal pain threshold | before chemotherapy & 3, 6, and 9 months after chemotherapy
  The threshold of detecting heat-induced pain

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No